# **Study protocol:**

| Title of study | Effects of Supervised Structured Aerobic Exercise training program on serum BDNF, |
|---|---|
| | androgens level, menstrual irregularity, aerobic fitness and quality of life in females |
| | with Insulin resistant polycystic ovarian syndrome. |
| Objective (s) of the | To determine the effects of Supervised Structured Aerobic Exercise Training |
| study | Program on quality of life in women with PCOS. |
| | 2. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on <b>BDNF levels</b> in women with PCOS. |
| | 3. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on mental health (stress, depression, anxiety) in women with PCOS. |
| | 4. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on <b>BMI</b> in women with PCOS. |
| | 5. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on menstrual irregularity in women with PCOS. |
| | 6. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on <b>Aerobic fitness</b> in women with PCOS. |
| | 7. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on androgens level in PCOS. |
| | 8. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on Lipid accumulation product in PCOS. |
| | 9. To determine the effect of Supervised Structured Aerobic Exercise Training |
| | Program on <b>Glycemic control</b> in PCOS. |
| Methodology | Design: RCT Randomized Controlled Trial |
| (Design samula | Non-probability Convenient Sampling Technique |
| (Design, sample | Duration of treatment: 25 weeks <b>2 groups</b> ; (group A=30) SSAET +Normal routine medication+ Normal Dietary Plan , Other |
| size, sampling | group (Group B=30) with normal routine medication + Normal Dietary Plan. |
| technique, Study | Patients will be enrolled in the experimental group according to speeds test. |
| setting, inclusion | |
| and exclusion | TOOLS |
| criteria and Tool) | TOOLS: 1. Modified polycystic ovarian syndrome Quality of Life Questionnaire |
| | (PCOSQOL)- Quality of life |
| | 2. MIQ (Menstrual Irregularity Questionnaire)- Menstrual irregularity |
| | 3. Women's weight in kilograms divided by the square of height in meters- BMI |
| | 4. A anahia fituasa |
| | 4. Aerobic fitness- |
| | YMCA 3-minute Bench Step Test, 3-Minute Step Test: |
| | You step up and down on a 30 cm (12-inch) step for three minutes at a |
| | consistent pace, and your heart rate is measured afterward to estimate |
| | fitness for 1 minute through carotid artery. The more fit you are, the |

lower your recovery heart rate will be, meaning a lower number is a better score.

# **Compare to Charts:**

Use your age and gender to find the appropriate fitness rating chart, such as the YMCA charts.

#### **Determine Your Level:**

The chart will show whether your 1-minute heart rate falls into categories like excellent, good, above average, average, or below average fitness.

# YMCA FEMALES Scoring:

Excellent < 109

Above Average 110 - 117

Average 118 - 134

Below Average 135-137

Poor >137

- 5. BDNF levels- ELISA
- 6. Androgens level- Serum SHBG will be measured by coated-tube immunoradiometric assay using commercial kits. Testosterone will be measured by RIA using commercial enzymatic kits. Free androgen index (FAI) will be calculated as testosterone/SHBG × 100.
  Clinical hyperandrogenism (a score of 6 or higher on the modified Ferriman–Gallwey scale)
- 7. **Mental health** (Stress, depression & Anxiety) by DASS-21 Severity Interpretation: Depression: The severity of depression is categorized as Normal (0-9), Mild (10-13), Moderate (14-20), Severe (21-27), and Extremely Severe (28+). Anxiety: The severity of anxiety is categorized as Normal (0-7), Mild (8-9), Moderate (10-14), Severe (15-19), and Extremely Severe (20+). Stress: The severity of stress is categorized as Normal (0-14), Mild (15-18), Moderate (19-25), Severe (26-33), and Extremely Severe (34+).
- 8. **Lipid Accumulation Product** -Triglycerides test and waist circumference The LAP would be calculated as [waist circumference (centimeters) – 58] × [triglycerides (millimoles per liter)]
- 9. Glycemic control- HOMA IR

The HOMA-IR score is calculated using your fasting glucose and fasting insulin levels:

HOMA-IR = (Fasting Glucose x Fasting Insulin) / 22.5

### **Rotterdum Criteria for a diagnosis of PCOS**

A diagnosis of PCOS can be made when at least two of the following three criteria are met:

1. Irregular periods or no periods

- 2. Higher levels of androgens are present in the blood (hyperandrogenism), shown by:
- a blood test, OR
- symptoms such as:
- o excess facial or body hair growth
- o scalp hair loss
- o acne.
- 3. Polycystic ovaries are visible on an ultrasound, meaning:
- more than 20 follicles (partly developed eggs) are visible on one or both ovaries or
- the size of one or both ovaries is increased (more than 10ml). You do not need to have an ultrasound if you have criteria 1 and 2.
- In women younger than 20 years, ultrasounds are not recommended. This means that irregular periods and hyperandrogenism need to be present for a diagnosis of PCOS to be made.

Study Setting: Gyms of Lahore

#### **Inclusion Criteria:**

- Age 18 To 35 years Females.
- Insuline resistant PCOS type.
- Already Diagnosed patients form gyne department according to the Rotterdam criteria.
- Both Married and unmarried females.
- Nulliparous females.

#### **Exclusion Criteria:**

- Post pill PCOS, Inflammatory PCOS & Adrenal PCOS
- Any psychological disease or disorder
- Any systemic disease other than PCOS (cushing syndrome, thyroid dysfunction, etc)
- Orthopedic conditions (including fracture, dislocation, etc)
- Any surgery in past 6 months.
- Involved in any other exercise regimen at the same time.
- Having any specialized diet plan.

\_

# Data analysis:

The data will be analysed using SPSS for Windows software, version 25. Statistical Significance will be set at P = 0.05. Normality of data will be assessed through Shapiro-Wilks test. Following tests will be used:

**Descriptive Statistics:** Frequency tables, pie charts, bar charts will be used to Show summary of group measurements measured over time.

# **Difference within groups:**

If the normality of data shows parametric result. Difference within group will be calculated using Repeated Measure ANOVA. For non-parametric data, Friedman test will be used.

# **Difference between Groups:**

Independent sample t test will be used for parametric data. If results are non-parametric then, then Mann Whitney U test will be used